CLINICAL TRIAL: NCT01971190
Title: Efficacy and Safety of Intravitreal Aflibercept Injection for Subacute Central Serous Chorioretinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young Hee Yoon, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFECT_001
Record Dates: First submitted 2013-10-21; First posted 2013-10-29 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham injection (Sham Comparator): Sham injection at baseline, at 1 month, and at 2 month
  Interventions: Drug: Sham injection; Procedure: Half-fluence photodynamic therapy
- Intravitreal Aflibercept injection (Active Comparator): 2mg intravitreal Aflibercept(Eylea) injection at baseline, at 1 month, and at 2 month
  Interventions: Drug: Intravitreal Aflibercept injection; Procedure: Half-fluence photodynamic therapy

INTERVENTIONS:
Drug: Intravitreal Aflibercept injection — 2mg intravitreal Aflibercept(Eylea) injection at baseline, at 1 month, and at 2 month.
  At 3 month, 4 month, 5 month, and 6 month, PRN treatment of aflibercept injection or half-fluence photodynamic therapy may be done, if one of following conditions is fulfilled.
  The PRN treatment method was decided by investigator's discretion.
  Of patient who had persistent intra- or subretina fluid on SD-OCT
  1. Central subfield thickness is not decreased to more than 50 micrometer compared with baseline central subfield thickness
  2. Best-corrected ETDRS letter score dose not increased more than 5 letters than baseline (because of the persistent CSC).
  3. Central subfield thickness is thicker than the previous exam
  4. BCVA letter score is worse than the previous exam (because of the persistent CSC)
  Arms: Intravitreal Aflibercept injection
Drug: Sham injection — Sham injection at baseline, at 1 month, and at 2 month.
  At 3 month, 4 month, 5 month, and 6 month, PRN treatment of aflibercept injection or half-fluence photodynamic therapy may be done, if one of following conditions is fulfilled.
  The PRN treatment method was decided by investigator's discretion.
  Of patient who had persistent intra- or subretina fluid on SD-OCT
  1. Central subfield thickness is not decreased to more than 50 micrometer compared with baseline central subfield thickness
  2. Best-corrected ETDRS letter score dose not increased more than 5 letters than baseline (because of the persistent CSC).
  3. Central subfield thickness is thicker than the previous exam
  4. BCVA letter score is worse than the previous exam (because of the persistent CSC)
  Arms: Sham injection
Procedure: Half-fluence photodynamic therapy — At 3 month, 4 month, 5 month, and 6 month, PRN treatment of aflibercept injection or half-fluence photodynamic therapy may be done, if one of following conditions is fulfilled.
  The PRN treatment method was decided by investigator's discretion.
  Of patient who had persistent intra- or subretina fluid on SD-OCT
  1. Central subfield thickness is not decreased to more than 50 micrometer compared with baseline central subfield thickness
  2. Best-corrected ETDRS letter score dose not increased more than 5 letters than baseline (because of the persistent CSC).
  3. Central subfield thickness is thicker than the previous exam
  4. BCVA letter score is worse than the previous exam (because of the persistent CSC)

SUMMARY:
Central serous chorioretinopathy (CSC) is a self-limiting disease that usually associated with good visual prognosis. In some cases, however, CSC may persist and result in permanent retinal or retinal pigment epithelium (RPE) damage. Therefore, if the disease is persistent beyond the acute phase, an active treatment should be considered to prevent an irreversible damage to retinal function.

The pathophysiology of CSC is associated with abnormal choroidal circulation. Indocyanine green angiography (ICGA) has revealed dilated and congested choroidal vessel and leakage into the extracellular space that appears as area of hyperfluorescence seen in middle and late phase in eyes with CSC.

A goal of treatment has been focused on reducing choroidal hyperpermeability. Currently, photodynamic therapy with verteporfin (PDT) and intravitreal anti-VEGF (vascular endothelial growth factor)antibody injection are being tried in order to treat chronic CSC. PDT reduces choroidal hyperpermeability by inducing hypoperfusion of the choriocapillaris in the short term and choroidal vascular remodeling over time. Intravitreal anti-VEGF injection for the treatment of CSC also effectively reduces choroidal hyperpermeability by blocking vascular leakage. Both methods have shown to be effective with good functional outcome for treating chronic CSC in many reports, but until now there is no established standard treatment protocol for chronic CSC.

Bevacizumab (Avastin) and ranibizumab (Lucentis) have been used widely as anti-VEGF therapeutic agent for the treatment of age related macular generation (AMD) and macular edema of various reasons. A newly developed anti-VEGF drug, aflibercept (Eylea○R), shows higher affinity to VEGF and has a longer duration of effect in the vitreous.FDA approved aflibercept to treat wet type AMD and macular edema due to central retinal vein occlusion.

Until now, no study has been reported on the efficacy and safety of aflibercept for treating CSC. The aim of this study is to evaluate the efficacy and safety of intravitreal aflibercept injection for the treatment of idiopathic CSC

DETAILED DESCRIPTION:
Single-center Double blind randomized Phase 2 interventional parallel study.

Group A : 2mg intravitreal Aflibercept(Eylea) injection at baseline, at 1 month, and at 2 month Group B : Sham injection at baseline, at 1 month, and at 2 month

At 3 month, 4 month, 5 month, and 6 month, PRN treatment of aflibercept injection or half-fluence photodynamic therapy may be done, if one of following conditions is fulfilled.

The PRN treatment method was decided by investigator's discretion.

Of patient who had persistent intra- or subretina fluid on SD-OCT

1. Central subfield thickness is not decreased to more than 50 micrometer compared with baseline central subfield thickness
2. Best-corrected ETDRS letter score dose not increased more than 5 letters than baseline (because of the persistent CSC).
3. Central subfield thickness is thicker than the previous exam
4. BCVA letter score is worse than the previous exam (because of the persistent CSC)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic CSC.
* 18 to 60 years old, woman and man.
* Subretinal fluid is found at OCT.
* Symptom duration is from 6 weeks to 4 months.
* Patient who agree to participate in the study.

Exclusion Criteria:

* Patient who was treated previously for CSC
* Patient who has choroidal neovascularization or other macular disease
* Patient who has other ophthalmologic disease that may affect patient's vision.
* History of any intraocular surgery, except cataract extraction prior to 3 months
* Patient who has active intraocular inflammation or infection
* Patient who has uncontrolled glaucoma IOP was more than 25 mmHg in spite of anti-glaucoma medication Visual field defect which affect best corrected visual acuity
* Patient who has been used systemic or topical carbonic anhydrase inhibitor within 1 month
* Cushing syndrome
* History of intravitreal steroid injection to study eye
* Patient who has been used or plan to use systemic drug which is toxic to crystalline lens, retina or optic nerve.
* Patient who has a known allergy to fluorescein or ICG
* Pregnant or breast-feeding woman
* Patient with contraindication to aflibercept Ocular or periocular infection Active severe intraocular inflammation Known hypersensitivity to aflibercept or to any of the excipients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes of central subfield thickness from baseline with time | at 1,2,3,4,5,6 month

SECONDARY OUTCOMES:
Percentage of eyes achieving complete resolution of subretinal fluid | at 6 month
Percentage of eyes achieving 20/20 vision | at 6 month
Number of aflibercept injection to achieve a complete resolution | at 6 month
Change in subfoveal choroidal thickness from baseline using EDI-OCT | at 1,2,3,4,5,6 month
Adverse effect of intravitreal aflibercept (Eylea) injection | upto 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Young Hee Yoon, MD, Principal Investigator — Asan Medical Center
Locations (6):
- South Korea (6):
  - Chungbuk national hospital, Chungju
  - Gangneung asan hospital, Gangneung
  - Seoul national university Bundang Hospital, Ilsan
  - Asan medical center, Seoul
  - Kim's Eye Hospital, Seoul
  - Samsung seoul hospital, Seoul

REFERENCES:
- [Background] Dohrmann J, Lommatzsch A, Spital G, Pauleikhoff D. [Pathogenesis of central serous chorioretinopathy: angiographic and electrophysiological studies]. Ophthalmologe. 2001 Nov;98(11):1069-73. doi: 10.1007/s003470170027. German. PMID 11729739
- [Background] Wong R, Chopdar A, Brown M. Five to 15 year follow-up of resolved idiopathic central serous chorioretinopathy. Eye (Lond). 2004 Mar;18(3):262-8. doi: 10.1038/sj.eye.6700637. PMID 15004575
- [Background] Spaide RF, Hall L, Haas A, Campeas L, Yannuzzi LA, Fisher YL, Guyer DR, Slakter JS, Sorenson JA, Orlock DA. Indocyanine green videoangiography of older patients with central serous chorioretinopathy. Retina. 1996;16(3):203-13. doi: 10.1097/00006982-199616030-00004. PMID 8789858
- [Background] Bae SH, Heo JW, Kim C, Kim TW, Lee JY, Song SJ, Park TK, Moon SW, Chung H. A randomized pilot study of low-fluence photodynamic therapy versus intravitreal ranibizumab for chronic central serous chorioretinopathy. Am J Ophthalmol. 2011 Nov;152(5):784-92.e2. doi: 10.1016/j.ajo.2011.04.008. Epub 2011 Jul 13. PMID 21742303
- [Background] Lee JY, Chae JB, Yang SJ, Kim JG, Yoon YH. Intravitreal bevacizumab versus the conventional protocol of photodynamic therapy for treatment of chronic central serous chorioretinopathy. Acta Ophthalmol. 2011 May;89(3):e293-4. doi: 10.1111/j.1755-3768.2009.01835.x. No abstract available. PMID 20346078
- [Background] Lim JW, Kim MU. The efficacy of intravitreal bevacizumab for idiopathic central serous chorioretinopathy. Graefes Arch Clin Exp Ophthalmol. 2011 Jul;249(7):969-74. doi: 10.1007/s00417-010-1581-9. Epub 2010 Dec 8. PMID 21140161
- [Background] Semeraro F, Romano MR, Danzi P, Morescalchi F, Costagliola C. Intravitreal bevacizumab versus low-fluence photodynamic therapy for treatment of chronic central serous chorioretinopathy. Jpn J Ophthalmol. 2012 Nov;56(6):608-12. doi: 10.1007/s10384-012-0162-3. Epub 2012 Aug 23. PMID 22915299
- [Background] Browning DJ, Kaiser PK, Rosenfeld PJ, Stewart MW. Aflibercept for age-related macular degeneration: a game-changer or quiet addition? Am J Ophthalmol. 2012 Aug;154(2):222-6. doi: 10.1016/j.ajo.2012.04.020. PMID 22813448
- [Background] Frampton JE. Aflibercept for intravitreal injection: in neovascular age-related macular degeneration. Drugs Aging. 2012 Oct;29(10):839-46. doi: 10.1007/s40266-012-0015-2. PMID 23038609
- [Background] Holash J, Davis S, Papadopoulos N, Croll SD, Ho L, Russell M, Boland P, Leidich R, Hylton D, Burova E, Ioffe E, Huang T, Radziejewski C, Bailey K, Fandl JP, Daly T, Wiegand SJ, Yancopoulos GD, Rudge JS. VEGF-Trap: a VEGF blocker with potent antitumor effects. Proc Natl Acad Sci U S A. 2002 Aug 20;99(17):11393-8. doi: 10.1073/pnas.172398299. Epub 2002 Aug 12. PMID 12177445
- [Background] Brown DM, Heier JS, Clark WL, Boyer DS, Vitti R, Berliner AJ, Zeitz O, Sandbrink R, Zhu X, Haller JA. Intravitreal aflibercept injection for macular edema secondary to central retinal vein occlusion: 1-year results from the phase 3 COPERNICUS study. Am J Ophthalmol. 2013 Mar;155(3):429-437.e7. doi: 10.1016/j.ajo.2012.09.026. Epub 2012 Dec 4. PMID 23218699
- [Background] Heier JS, Brown DM, Chong V, Korobelnik JF, Kaiser PK, Nguyen QD, Kirchhof B, Ho A, Ogura Y, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Soo Y, Anderesi M, Groetzbach G, Sommerauer B, Sandbrink R, Simader C, Schmidt-Erfurth U; VIEW 1 and VIEW 2 Study Groups. Intravitreal aflibercept (VEGF trap-eye) in wet age-related macular degeneration. Ophthalmology. 2012 Dec;119(12):2537-48. doi: 10.1016/j.ophtha.2012.09.006. Epub 2012 Oct 17. PMID 23084240
- [Background] Boyer D, Heier J, Brown DM, Clark WL, Vitti R, Berliner AJ, Groetzbach G, Zeitz O, Sandbrink R, Zhu X, Beckmann K, Haller JA. Vascular endothelial growth factor Trap-Eye for macular edema secondary to central retinal vein occlusion: six-month results of the phase 3 COPERNICUS study. Ophthalmology. 2012 May;119(5):1024-32. doi: 10.1016/j.ophtha.2012.01.042. Epub 2012 Mar 21. PMID 22440275
- [Background] Do DV, Nguyen QD, Boyer D, Schmidt-Erfurth U, Brown DM, Vitti R, Berliner AJ, Gao B, Zeitz O, Ruckert R, Schmelter T, Sandbrink R, Heier JS; da Vinci Study Group. One-year outcomes of the da Vinci Study of VEGF Trap-Eye in eyes with diabetic macular edema. Ophthalmology. 2012 Aug;119(8):1658-65. doi: 10.1016/j.ophtha.2012.02.010. Epub 2012 Apr 24. PMID 22537617
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203